CLINICAL TRIAL: NCT06320925
Title: A Retrospective, Multi-Center, Post-Market Clinical Follow-Up Study of Stryker Class IIb Implants
Brief Title: SportsPro: Post-Market Clinical Follow Up Study
Status: Recruiting | Type: Observational
Sponsor: Stryker Endoscopy (Industry)
Responsible Party: Sponsor
Other Study IDs: SYK-SM-2022-02
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Injuries; Knee Injuries; Hip Injuries
MeSH Terms: conditions — Shoulder Injuries; Knee Injuries; Hip Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Subjects: Patients who have undergone a surgical procedure (per product indications for use) using the Stryker implants who meet all of the following criteria will be screened and enrolled by participating Investigators.
  Interventions: Device: Standard of Care Treatment

INTERVENTIONS:
Device: Standard of Care Treatment — Subject has undergone joint space repair using one of the study devices and meets eligibility criteria

SUMMARY:
Retrospective, multi-center, chart review (only to include data that is part of the surgeons' standard practice)

DETAILED DESCRIPTION:
The purpose of this study is to leverage standard of care data to provide further characterization of clinical outcomes following shoulder, hip and knee joint surgeries.

* Primary Objective: To describe clinical outcomes of the Stryker Device in the shoulder, hip, and knee joints 6 months after surgical intervention.
* Secondary Objective: To describe clinical outcomes of the Stryker Device in the shoulder, hip, and knee joints 3 months after surgical intervention.
* Safety Objective: To describe safety of the Stryker implants in the shoulder, hip, and knee joints 6 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was ≥ 18 years of age at the time of the surgery
2. Subject has undergone joint space repair using one of the study devices

Exclusion Criteria:

1. Subjects who are less than 6 months post-intervention
2. Concurrent participation in an investigational clinical study during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone a surgical procedure (per indications for use) using the Stryker implants who meet all of the inclusion/exclusion criteria will be screened and enrolled by participating Investigators.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
ASES | 6 months
  Change from baseline
iHOT-12 | 6 months
  Change from baseline
mHHS | 6 months
  Change from baseline

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Musculoskeletal-Orthopedic Research and Education Foundation, Phoenix, Arizona
  - Steadman Hawkins Clinic Denver, Englewood, Colorado
  - TSAOG Orthopaedics & Spine, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No